CLINICAL TRIAL: NCT02007668
Title: Is Kinesio Taping More Effective Than Medical Adhesive Tape in Patients With Chronic Non-specific Low Back Pain? A Randomized Controlled Trial
Brief Title: Is Kinesio Taping More Effective Than Medical Adhesive Tape in Patients With Chronic Non-specific Low Back Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Mauricio Antonio da Luz Junior, Kinesio Taping is More Effective Than Medical Adhesive Tape in Patients With Chronic Non-specific Low Back Pain? A Randomized Controlled Trial, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE:16832013.9.0000.5512
Record Dates: First submitted 2013-11-30; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Low Back Pain
Keywords: low back pain; kinesio taping
MeSH Terms: conditions — Low Back Pain | interventions — Bandages; Athletic Tape

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio Taping (Experimental): Patients will receive an application of Kinesio taping in their lumbar spine.
  Interventions: Other: Kinesio Taping
- Kinesio Taping Placebo (Placebo Comparator): Patients will receive an application of medical adhesive tape in their lumbar spine.
- Control (No Intervention): This participants will not receive intervention

INTERVENTIONS:
Other: Kinesio Taping — Kinesio taping intervention is based upon the use of specific elastic tapes (known as Kinesio Tex Gold) that are applied with a certain amount of tension fixed to the skin of patients with the target muscles in a stretched position. The tapes will be placed over the lumbar spine.
  Other Names: -Bandages; -Tape; -Taping; -Kinesio Tex; -Kinesio Tape; -Kinesiotape
  Arms: Kinesio Taping

SUMMARY:
Sixty patients will be randomized into three groups to receive the Kinesio taping, placebo Kinesio taping (medical adhesive tape) and control group. The group Kinesio taping receive the correct application of the method described. The placebo group will receive a medical adhesive tape. The control group will not receive any form of intervention.

DETAILED DESCRIPTION:
The group Kinesio taping receive the correct application of the method described with tension paper off (10-15%). The placebo group will receive a medical adhesive tape. The control group will not receive any form of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific low back pain longer than 3 months
* Seeking care for low back pain

Exclusion Criteria:

* Contra indications to any bandage
* Serious sinal pathologies (e.g. tumors, fractures and inflammatory diseases)
* Nerve roto compromise
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 2 days
  Pain Intensity will be measured in 2 and 7 days after randomization by an 11-point (0-10) Numerical Rating Scale (Pain NRS)

SECONDARY OUTCOMES:
Disability | 2 days
  Disability associated with low back pain will be measured in 2 and 7 days after randomization by the 24-item Roland Morris Disability Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Antonio da Luz Junior, MSc, Principal Investigator — Paulista University
Locations (1):
- Universidade Paulista - UNIP, Jundiaí, São Paulo, Brazil